CLINICAL TRIAL: NCT04163835
Title: The Dose-Effect Relationship of Wenxin Granules in the Treatment of Atrial Premature Beats of Deficiency of Both Qi and Yin and Heart Vessel Stasis and Obstruction Syndrome : A Randomized, Double-blind, Placebo-controlled Clinical Trial Study
Brief Title: The Dose-Effect Relationship of Wenxin Granules in the Treatment of Atrial Premature Beats
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WX20150820
Record Dates: First submitted 2019-10-29; First posted 2019-11-15 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Atrial Premature Complexes
Keywords: Wenxin Granules; Dose-effect relationship; Deficiency of both Qi and Yin Syndrome; Heart Vessel Stasis and Obstruction Syndrome; Traditional Chinese Medicine; arrhythmia
MeSH Terms: conditions — Atrial Premature Complexes; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: The ratio of high, medium and low dose group and placebo groups are 1:1:1:1. A total of 60 cases are included in the first phase.The maximum sample size required is determined to be 150 cases.
Who Masked: Participant, Investigator
Masking Description: This study was a double-blind clinical trial, with the patients, the treating physicians, the statisticians, the monitors and any other personnel being unaware of group allocation. Efforts to maintain blinding included identical appearance, packaging and labeling of four groups of experimental drugs.
  Unblinding should be done by the statisticians when the data collection process was completed or the treating physicians when serious adverse events occurred.
  The maximum sample size required is determined to be 150 cases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-dose Group (Experimental): The intervention is half-dose of Wenxin Granules (1/2 normal dose).
  Interventions: Drug: 1/2 Normal-dose Wenxin Granules
- Medium-dose Group (Experimental): The intervention is medium-dose of Wenxin Granules (normal dose).
  Interventions: Drug: Normal-dose Wenxin Granules
- High-dose Group (Experimental): The intervention is twice-dose of Wenxin Granules (twice normal dose).
  Interventions: Drug: Twice Normal-dose Wenxin Granules
- Placebo Group (Placebo Comparator): The intervention is a placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Normal-dose Wenxin Granules — The drugs should be taken 10 g orally each time, 3 times a day after meals, for 4 weeks.
  Ingredients: Wenxin Granules (no sucrose) 5g + Wenxin Granules placebo 5g.
  Arms: Medium-dose Group
Drug: 1/2 Normal-dose Wenxin Granules — The drugs should be taken 10 g orally each time, 3 times a day after meals, for 4 weeks.
  Ingredients: Wenxin Granules (no sucrose) 2.5g + Wenxin Granules placebo 7.5g.
  Arms: Low-dose Group
Drug: Twice Normal-dose Wenxin Granules — The drugs should be taken 10 g orally each time, 3 times a day after meals, for 4 weeks.
  Ingredients: Wenxin Granules (no sucrose) 10g.
  Arms: High-dose Group
Drug: Placebo — The drugs should be taken 10 g orally each time, 3 times a day after meals, for 4 weeks.
  Ingredients: Wenxin Granules placebo 10g.
  Arms: Placebo Group

SUMMARY:
A Randomized, double-blind, placebo-controlled, four dose groups, post-marketing clinical trial, to evaluate the efficacy and safety of Wenxin granules in treating atrial premature beats by different doses,to provide a scientific basis for rational clinical use of drug.

DETAILED DESCRIPTION:
Research purpose: To evaluate the efficacy and safety of Wenxin granules in treating atrial premature beats by different doses, to provide a scientific basis for rational clinical use of drug.

Research design: A Randomized, double-blind, placebo-controlled, four dose groups, post-marketing clinical trial.

Sample size:

The ratio of high, medium and low dose groups and placebo group were 1:1:1:1. A total of 60 cases were included in the first phase.The maximum sample size required was determined to be 150 cases.

Therapeutic schedule:

1. Low-dose Group(1/2 Normal-dose Wenxin Granules ):Wenxin Granules (no sucrose) 2.5g + Wenxin Granules placebo 7.5g.
2. Medium-dose Group(Normal-dose Wenxin Granules ):Wenxin Granules (no sucrose) 5g + Wenxin Granules placebo 5g.
3. High-dose Group(Twice Normal-dose Wenxin Granules):Wenxin Granules (no sucrose) 10g.
4. Placebo Group(Placebo):Wenxin Granules placebo 10g.

Usage and Dosage:The drugs should be taken 10 g orally each time, 3 times a day after meals, for 4 weeks.

Drug combination:

During the test should not merge the other anti-arrhythmic drugs beyond the provisions of this scheme. Due to merger disease or condition changes ,have to use drugs or other treatment, investigators must record the types (or other treatment ),drug usage, time and reasons, in order to summarize ,analyze and report.

Primary Outcome Measures

1. Responder rate based on 24-hour Holter monitoring, defined as the proportion (%) of subjects with a ≥ 50% reduction in atrial premature beats during 24-hour Holter monitoring from baseline.

Time Frame: Week 0 to Week 4

Secondary Outcome Measures

1. Change in Total Score From Baseline in Traditional Chinese Medicine Syndrome Score Scale (TCMSSS).

   Time Frame: Week 0 to Week 4
2. Responder rate based on each symptom score, defined as the proportion (%) of subjects with a ≥ 1 score reduction in each symptom score from baseline.

Time Frame: Week 0 to Week 4

Other Outcome Measures

1. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 Time Frame: Week 0 to Week 4
2. Impact of treatment on Liver Function Time Frame: Week 0 to Week 4
3. Impact of treatment on Renal Function Time Frame: Week 0 to Week 4
4. Impact of treatment on Hemoglobin Levels Time Frame: Week 0 to Week 4
5. Impact of treatment on White Blood Cells Time Frame: Week 0 to Week 4
6. Impact of treatment on Blood Platelet Time Frame: Week 0 to Week 4
7. Impact of treatment on Hematuria and Proteinuria Time Frame: Week 0 to Week 4

ELIGIBILITY:
Inclusion Criteria:

1. Accord with the diagnostic criteria of arrhythmia (atrial premature beats );
2. Accord with the diagnostic criteria of deficiency of both qi and yin and heart vessel stasis and obstruction Syndrome;
3. The number of premature beat of 24 h dynamic electrocardiogram >360 times/h or >8640 times/24h;
4. Stop using the anti- arrhythmic drugs for more than five half-life (except that who long-term (one month or more) with beta blockers for high blood pressure and exertional angina);
5. Ages 18 to 75 years old ,all genders;
6. Voluntary subjects and signed the informed consent form.

Exclusion Criteria:

1. Serious condition that need to merge other anti-arrhythmic drugs(I,II,III,IV) to treat;
2. Heart rhythm disorders caused by the factors such as drugs ,electrolyte and acid-base balance disorders;
3. Merge tardy arrhythmia (including sick sinus syndrome and II degree atrioventricular block);
4. Removed predisposing factors (such as fatigue, nervousness, mood swings, alcoholism, etc.) the premature beats reduced, while the symptoms significantly relieved;
5. Patients who have pacemaker implanted or have undergone heart percutaneous coronary intervention (PCI) surgery;
6. Patients with severe hypotension;
7. Patients with serious cardiovascular diseases (such as congestive heart failure, cardiac shock, etc.), cerebrovascular disease, and serious primary 8.diseases such as liver, kidney and hematopoietic system (ALT,AST,BUN 2 times higher than normal ceiling, or Cr higher than the upper limit of normal);
8. Allergic constitution; the test drug allergy or its ingredients or elements allergy;
9. Pregnancy and lactation women ,recent preparation pregnancy;
10. Patients with chronic alcoholism , drug dependence, mental illness;
11. Participated in other clinical trials within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Responder rate based on 24-hour Holter monitoring. | Week 0 to Week 4
  Defined as the proportion (%) of subjects with a ≥ 50% reduction in atrial premature beats during 24-hour Holter monitoring from baseline.

SECONDARY OUTCOMES:
Change in Total Score From Baseline in Traditional Chinese Medicine Syndrome Score Scale. | Week 0 to Week 4
  The rating scale consisted of 12 items (1 for the main symptoms and 11 for the accompanying symptoms) with 4 options (absent, mild, moderate or severe) for each item. Each option was represented by a fixed score(0,1,2,3), the higher the score, the more severe the symptom, and vice versa. The total score of the rating scale was called syndrome integral.
  Symptoms include palpitation, chest distress, chest pain, shortness of breath, lack of strength, insomnia, dreamfulness, dizziness, dim complexion, vexing heat in chest, palms and soles, dry mouth, cyanotic lips and nails.
  The changes of TCM syndrome scores before and after treatment were compared.
Responder rate(%) based on each symptom score. | Week 0 to Week 4
  Defined as the proportion (%) of subjects with a ≥ 1 score reduction in each symptom score from baseline.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Week 0 to Week 4
  Following drug administration, a review of subjective symptoms will be performed.
Impact of treatment on Liver Function | Week 0 to Week 4
  Blood samples will be collected to examine the impact of treatment on the levels of ALT, AST in the subjects blood.
Impact of treatment on Renal Function | Week 0 to Week 4
  Blood samples will be collected to examine the impact of treatment on the levels of Cr, Bun in the subjects blood.
Impact of treatment on Hemoglobin Levels | Week 0 to Week 4
  Blood samples will be collected to examine the impact of treatment on the levels of Hemoglobin in the subjects blood.
Impact of treatment on White Blood Cells | Week 0 to Week 4
  Blood samples will be collected to examine the impact of treatment on the levels of white blood count in subjects blood.
Impact of treatment on Blood Platelet | Week 0 to Week 4
  Blood samples will be collected to examine the impact of treatment on the levels of Blood Platelet in subjects blood.
Impact of treatment on Hematuria and Proteinuria | Week 0 to Week 4
  Urine samples will be collected to examine the the presence and amount of blood and protein in the urine.

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Wu, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No